CLINICAL TRIAL: NCT04231942
Title: Elastic Compression Stockings in the Prevention of Varicose Veins Recurrence After Endovenous Thermal Ablation
Brief Title: Elastic Compression Stockings and Varicose Veins Recurrence
Acronym: ECOS-VVR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECOS-VVR
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Varicose Veins; Chronic Venous Insufficiency
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Intervention Model Description: A multicenter, open, superiority randomized clinical trial with blinded outcome assessor.
Who Masked: Outcomes Assessor
Masking Description: Blinded outcome assessor has np information on the patients belonging to the Study Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (experimental): continuous using of GCS (Experimental): At 30-45 days after the intervention for VVs treatment patients without objective signs (C0-1) and subjective symptoms (intensity of 30% and less) of CVD, without any need for long-term using of GCS and/or vein-active drugs will receive appropriate recommendations on lifestyle correction (avoiding long static activities, maintaining an active lifestyle, the correction of excess weight and constipation, a diet with enough fiber and vitamins) and physical activity (visiting the pool, exercises that improve venous outflow).
  In addition to lifestyle correction and exercises, patients will be recommended to use Class 1 (RAL GZ 387) below-knee GCS (at least 8 hours per day) for both lower extremities every day for 12 months, while change of GCS for the new one should be carried out at 6 months or early in case of stocking deterioration;
  Interventions: Device: Graduated Compression Stocking: continuous using
- Group 2 (experimental): intermittent using of GCS (Experimental): At 30-45 days after the intervention for VVs treatment patients without objective signs (C0-1) and subjective symptoms (intensity of 30% and less) of CVD, without any need for long-term using of GCS and/or vein-active drugs will receive appropriate recommendations on lifestyle correction (avoiding long static activities, maintaining an active lifestyle, the correction of excess weight and constipation, a diet with enough fiber and vitamins) and physical activity (visiting the pool, exercises that improve venous outflow).
  In addition to lifestyle correction and exercises, patients will be recommended to use Class 1 (RAL GZ 387) below-knee GCS on both limbs during physical activity and long stasis events: any kind of sport activities, air travel of any duration, traveling on vehicles for more than 4 hours, walking for more than 2 hours, standing work for more than 4 hours) for 12 months, while change of GCS for the new one should be carried in case of stocking deterioration;
  Interventions: Device: Graduated Compression Stocking: intermittent using
- Group 3 (control): no use of GCS (No Intervention): At 30-45 days after the intervention for VVs treatment patients without objective signs (C0-1) and subjective symptoms (intensity of 30% and less) of CVD, without any need for long-term using of GCS and/or vein-active drugs will receive appropriate recommendations on lifestyle correction (avoiding long static activities, maintaining an active lifestyle, the correction of excess weight and constipation, a diet with enough fiber and vitamins) and physical activity (visiting the pool, exercises that improve venous outflow).
  The use of GCS will be possible "on-demand" when symptoms or risk factors appear after appropriate coordination with the Investigator

INTERVENTIONS:
Device: Graduated Compression Stocking: continuous using — Class 1 (RAL-GZ 387 standard: 18-21 mm Hg at the ankle level) below-knee graduated compression stockings
  Arms: Group 1 (experimental): continuous using of GCS
Device: Graduated Compression Stocking: intermittent using — Class 1 (RAL-GZ 387 standard: 18-21 mm Hg at the ankle level) below-knee graduated compression stockings
  Arms: Group 2 (experimental): intermittent using of GCS

SUMMARY:
Hypothesis. Regular using of Class 1 below-knee graduated compression stockings (RAL GZ 387 standard) compared to the absence of elastic compression will reduce the risk of clinically significant varicose veins recurrence at 12 months after endovenous thermal ablation of the great saphenous vein and elimination of varicose tributaries.

DETAILED DESCRIPTION:
The incidence of new varicose veins (VVs) appearance at 3 years after any invasive treatment is about 20%, and the progression rate of chronic venous disease (CVD) at 2 years after the endovenous thermal ablation (ETA) reaches 40%. When comparing open surgery and endovenous laser ablation (EVLA), the frequency of VVs recurrence at 12 months after intervention does not significantly differ and amounts to 10%. A previous study examining the effect of elastic compression on the risk of VVs recurrence after surgery showed a 92% reduction in relative risk. However, it was limited to the low number of followed patients and the absence of the compliance measurement. Thus, there is still no evidence, if long term using of graduated compression stockings (GSV) after modern modalities of VVs treatment (ETA with mini/micro phlebectomy or sclerotherapy) provides any benefits in the reduction of VVs recurrence. Also, there is no information on what regimen for GCS using is effective to reduce the risk of VVs recurrence: continuous use at every day or intermittent using only during specific activities.

Our hypothesis is that regular using of Class 1 below-knee graduated compression stockings (RAL GZ 387 standard) compared to the absence of elastic compression will reduce the risk of clinically significant varicose veins recurrence at 12 months after endovenous thermal ablation of the great saphenous vein and elimination of varicose tributaries.

The aim of the study is to assess the efficacy of regular using of below-knee graduated compression stockings (GCS) of Class 1 (RAL-GZ 387 standard: 18-21 mm Hg at the ankle level) on the risk of varicose veins clinical recurrence after endovenous thermal obliteration of the great saphenous vein and eliminating varicose tributaries in patients without residual varicose veins and / or venous symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Varicose veins (VVs) in the system of great saphenous vein (GSV) of one lower limb;
* Performed endovenous thermal ablation (ETA) of the GSV trunk - endovenous laser ablation (EVLA) or radiofrequency ablation (RFA) - and elimination of varicose tributaries by mini (micro) phlebectomy or sclerotherapy during the 30-45 days before enrollment;
* The technical success of the performed ETA, the absence of reflux in the GSV trunk and the absence of residual VVs;
* Lack of signs of chronic venous disease (CVD): clinical class of C0-1 according to the Clinical-Etiology-Anatomy-Pathophysiology (CEAP) classification;
* Lack of vein-specific symptoms - the intensity of any validated vein-specific symptom is less than 30% according to the numeric rating scale (NRS);
* Signed informed consent.

Exclusion Criteria:

* Bilateral VVs;
* Primary reflux outside the GSV trunk (including combined);
* History of deep or superficial veins thrombosis;
* Verified deep vein reflux;
* Verified non-thrombotic or post-thrombotic venous obstruction;
* Verified pelvic venous insufficiency;
* Persistence of superficial reflux after ETA;
* A tendency for recanalization of previously obliterated veins;
* Persistence of residual VVs - clinical class of C2 by CEAP;
* Persistence of signs of CVD - clinical class of C3 and higher by CEAP;
* Persistence of one or more vein-specific symptom with an intensity of 30% and higher by NRS;
* The need for long-term use of elastic compression;
* Contraindications or restrictions for the long-term use of GCS;
* The need for long-term use of vein-active drugs (more than 1 month);
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with clinical recurrence of varicose veins on any lower limb | 12 months
  The primary efficacy outcome is the clinical recurrence of varicose veins at 12 months after the treatment, which means the reappearance of the visible or palpable varicose tributaries on any (treated or non-treated) lower limb.

SECONDARY OUTCOMES:
Number of patients with clinical recurrence of varicose veins on treated limb | 12 months
  The reappearance of the visible or palpable varicose tributaries on treated lower limb
Number of patients with ultrasound recurrence of varicose veins on any lower limb | 12 months
  The appearance of invisible and non-palpable VVs on any (treated or non-treated) limb revealed by duplex ultrasound scan (DUS)
Number of patients with ultrasound recurrence of varicose veins on treated limb | 12 months
  The appearance of invisible and non-palpable VVs on treated lower limb revealed by duplex ultrasound scan
Number of patients with recanalization of obliterated great saphenous vein | 12 months
  The venous segment of the previously obliterated great saphenous vein (GSV) with blood flow revealed by DUS and the length of 5 cm and more
Number of patients underwent re-intervention for VVs | 12 months
  Any re-intervention to treat new varicose veins on treated or non-treated lower limb
Number of patients with C0-C1 clinical classes of СVD by CEAP classification | 12 months
  Clinical-Etiology-Anatomy-Pathophysiology (CEAP) classification of the chronic venous disease (CVD). Clinical class of C0 - no visible changes; Clinical class of C1- reticular veins and telangiectasia
The value of VCSS on the treated limb | 12 months
  The severity of CVD in the target lower limb is assessed during clinical examination using the updated Venous Clinical Severity Score (VCSS). Ranges from 0 to 30. Maximal score indicates more severe CVD.
The value of CIVIQ-20 score | 12 months
  The quality of life is assessed by the patient independently according to the vein-specific questionnaire Chronic Lower Limb Venous Insufficiency Questionnaire - 20 items (CIVIQ-20). range 0-100, minimal score indicates best quality of life.
Compliance with the use of GCS | 12 months
  Compliance with the use of GCS is assessed based on an analysis of the patient's individual diary. For Group 1 and 2, it is calculated as the ratio of days with a note on the using of GCS to the total number of days when compression is recommended: for Group 1 - the total observation period, for Group 2 - days with indicated activities. For Group 3, compliance is calculated as the total number of days of GCS using to the observation period. Ranges from 0% (no compliance) to 100% (absolute compliance).
Comfort with GCS | 12 months
  Comfort with GCS using is assessed individually by patient by Numeric Rating Scale (NRS). Ranges from 0 (no comfort) to 100% (absolute comfort).

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Laberko, PhD, Study Chair — Pirogov RNRMU; Leonid Laberko, PhD, Principal Investigator — Pirogov RNRMU
Locations (3):
- Russia (3):
  - Moscow Clinical Hospital name by A.K. Yeramishantsev, Moscow
  - Moscow Clinical Hospital no.24, Moscow
  - Moscow private medical clinic "MedSwiss", Moscow

IPD SHARING:
Plan to Share IPD: No